CLINICAL TRIAL: NCT01060254
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Explore the Efficacy, Safety, and Tolerability of JNJ-42160443 in Subjects With Interstitial Cystitis/ Painful Bladder Syndrome
Brief Title: A Study to Evaluate the Pain Relieving Effects, Safety, and Tolerability of JNJ-42160443 for the Relief of Bladder Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Logistic reasons associated with the FDA-imposed clinical hold.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR017017; 42160443PAI2005 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.); 2009-009856-19 (EudraCT Number: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Cystitis, Interstitial; Urologic Diseases; Urinary Bladder Diseases; Cystitis
Keywords: Interstitial cystitis (IC) and/or painful bladder syndrome (PBS)-related pain; Moderate to severe chronic bladder pain; JNJ-42160443
MeSH Terms: conditions — Cystitis, Interstitial; Urologic Diseases; Urinary Bladder Diseases; Cystitis | interventions — fulranumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- JNJ-42160443 (Experimental)
  Interventions: Drug: JNJ-42160443
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Form=solution for injection, route=Subcutaneous injection. One injection of matching placebo every 28 days for up to 12 wks
  Arms: Placebo
Drug: JNJ-42160443 — Type=exact number, unit=mg, number= 9, form=solution for injection, route=Subcutaneous use. One injection of 9 mg of JNJ-42160443 every 28 days for up to 12 wks
  Arms: JNJ-42160443

SUMMARY:
The purpose of this study is to evaluate the analgesic efficacy, safety, and tolerability of JNJ-42160443 compared to placebo in patients with moderate to severe, chronic bladder pain from interstitial cystitis and/or painful bladder syndrome.

DETAILED DESCRIPTION:
This study is a randomized (study drug assigned by chance), double-blind (neither the physician nor the patient knows the name of the assigned drug) study to evaluate the analgesic efficacy, safety, and tolerability of JNJ-42160443 compared with placebo in patients with moderate to severe, chronic bladder pain from Interstitial cystitis (IC) and/or painful bladder syndrome (PBS). Interstitial cystitis (IC) and PBS are urological disorders characterized by symptoms of bladder pain, urinary urgency, urinary frequency, and the need to get up during the night in order to urinate. The study has 3 phases: a screening phase (up to 3 weeks), a double-blind treatment phase (12 weeks), and a post-treatment phase that ends 26 weeks after the last dose of study medication. The study duration will be approximately 36 to 46 weeks.

A single dose of JNJ-42160443 (9 mg/ml) or matching placebo given as an injection under the skin once every 4 weeks for up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pelvic pain (>6 months) perceived to be related to the urinary bladder and accompanied by urinary symptoms such as frequent urination during the day and/or night, and/or urgency to void
* Total score of 8 or greater on the O'Leary-Sant Interstitial Cystitis Symptom Index (ICSI)
* The mean of the average pain intensity scores at screening phase >=5 (on a scale of 0 to 10)
* Medically stable

Exclusion Criteria:

* Urinary culture is positive for a urinary tract infection; Recent invasive therapy to the bladder
* History or current conditions indicating that the bladder pain can be caused by diagnoses other than IC/PBS (eg, pain caused by a confirmed or suspected neoplasm)
* History of malignancy within the past 2 years, with the exception of basal cell carcinoma that has been successfully treated
* Women who are pregnant or breast-feeding
* A body mass index (BMI) of >39 kg/m2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-04-06 (Actual); Primary Completion 2011-06-24 (Actual); Study Completion 2011-06-24 (Actual)

PRIMARY OUTCOMES:
The change in the average pain intensity score. | The change from baseline to the end of the double-blind phase in the mean average pain intensity score (12 weeks).

SECONDARY OUTCOMES:
Evaluation of Global Response Assessment (GRA) | 12 weeks
Changes from baseline in O'Leary-Sant Interstitial Cystitis Symptom Index (ICSI) | 12 weeks
Change in Pelvic Pain and Urgency/Frequency Questionnaire (PUF) | 12 weeks
Changes from baseline to end of the double-blind phase in subscale scores of the Short Form (SF)-12 Health Survey | 12 weeks
Antibody against JNJ-42160443 | 34 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (25):
- United States (20):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Glendora, California
  - San Diego, California
  - Aventura, Florida
  - Eagle, Idaho
  - Jeffersonville, Indiana
  - Kansas City, Kansas
  - Overland Park, Kansas
  - Metairie, Louisiana
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Brighton, Massachusetts
  - Royal Oak, Michigan
  - Englewood, New Jersey
  - Poughkeepsie, New York
  - Greensboro, North Carolina
  - Winston-Salem, North Carolina
  - Arlington, Texas
  - Fair Oaks Ranch, Texas
- Canada (5):
  - Barrie, Ontario
  - Kingston, Ontario
  - Kitchener, Ontario
  - North York, Ontario
  - Toronto, Ontario

REFERENCES:
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597
- [Derived] Wang H, Russell LJ, Kelly KM, Wang S, Thipphawong J. Fulranumab in patients with interstitial cystitis/bladder pain syndrome: observations from a randomized, double-blind, placebo-controlled study. BMC Urol. 2017 Jan 5;17(1):2. doi: 10.1186/s12894-016-0193-z. PMID 28056917